CLINICAL TRIAL: NCT06408597
Title: The Use of Intra-operative Mannitol Versus Nitroglycerin to Prevent Post-operative Acute Kidney Injury in Patients Undergoing Robotic-assisted Radical Prostatectomy or Cystectomy: A Randomized Controlled Trial.
Brief Title: Mannitol Versus Nitroglycerin for Kidney Injury Prevention in Robotic-assisted Radical Prostatectomy or Cystectomy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nazmy Edward Seif (Other)
Responsible Party: Sponsor-Investigator, Nazmy Edward Seif, Clinical Professor, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MVTKIPRARPC
Record Dates: First submitted 2024-05-07; First posted 2024-05-10 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Prostate Cancer; Bladder Cancer; Surgery; Renal Impairment; Renal Injury, Acute
Keywords: Radical Prostatectomy; Radical Cystectomy; Robotic; Anesthesia; Mannitol; Nitroglycerin
MeSH Terms: conditions — Prostatic Neoplasms; Urinary Bladder Neoplasms; Renal Insufficiency; Acute Kidney Injury

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Active Comparator): Standard Fluid Therapy group
  Interventions: Procedure: Fluid Regimen
- Nitroglycerin group (Experimental): Nitroglycerin Infusion group
  Interventions: Procedure: Nitroglycerin Infusion; Procedure: Fluid Regimen
- Mannitol group (Experimental): Mannitol Infusion group
  Interventions: Procedure: Mannitol Infusion; Procedure: Fluid Regimen

INTERVENTIONS:
Procedure: Nitroglycerin Infusion — Nitroglycerin prepared using a vial (50 mg nitroglycerin) transferred into a 500 ml glass bottle of sodium chloride injection (0.9%), this yields a concentration of 100 mcg/ml.
  Patients in the nitroglycerin group will receive nitroglycerin infusion at a rate of 0.25 mic/kg/min all through the surgery, to be discontinued in the PACU.
  Arms: Nitroglycerin group
Procedure: Mannitol Infusion — Mannitol will be prepared through diluting 100 ml of the 20% solution with 180 ml of sodium chloride injection (0.9%).
  Patients in the mannitol group will receive an infusion bolus of mannitol 20% 0.5gm/kg added to the standard fluid chart via centeral line.
  Mannitol intake will be started directly after induction of anaesthesia and before intra-peritoneal gas insufflation, as an infusion over 15 minutes.
  Arms: Mannitol group
Procedure: Fluid Regimen — Patients will take the standard fluid chart, as the patient will receive the estimated maintenance & deficit requirements according to 4/2/1 rule.
  In case of hypotension, (defined as 20% decrease from the baseline), administration of a fluid bolus of 200 ml ringer will be done.
  Blood loss more than 10% of estimated blood volume will initiate blood transfusion using 1:1 ratio. Additional fluids may be administered postoperatively according to the patient's volume status.

SUMMARY:
Laparoscopic and minimally-invasive robotic access has transformed the delivery of urological surgery. While associated with numerous desirable outcomes including shorter post-operative stay and faster return to preoperative function, these techniques have also been associated with morbidity such as reduced renal blood flow and post-operative renal dysfunction. The mechanisms leading to these renal effects complex are multifactorial, and have not been fully elucidated. However they are likely to include direct effects from raised intra-abdominal pressure, and indirect effects secondary to carbon dioxide absorption, neuroendocrine factors and tissue damage from oxidative stress. It is well documented that pneumoperitoneum places profound stress on the cardiovascular, respiratory and gastrointestinal systems; it also places strain on the renal system.

During robotic surgery, continuous pneumoperitoneum and continuous rising of intra-abdominal pressure causes transient oliguria. Moreover, kidney function, estimated by the GFR, deteriorates during elevated intra abdominal pressure (IAP), and most of the studies identified decrease in renal blood flow (RBF) and renal cortical perfusion.

Studies conducted to assess the contribution of the nitric oxide (NO) system to the renal hemodynamic/function alterations during pneumoperitoneum, concluded that these adverse effects are probably related to interference with the NO system, and could be partially ameliorated by pretreatment with nitroglycerine.

Mannitol is an osmotic diuretic and a renal vasodilator that promotes tubular flow, prevents intratubular cast formation, decreases postischemic cellular swelling, and might serve as a free radical scavenger. Mannitol has traditionally been administered before renal surgeries to minimize perioperative renal dysfunction according to preclinical animal studies and clinical experience with renal transplantation. However, high-level clinical data in support of this belief are not available.

The aim of this study is to characterize the effects of increased intra-abdominal pressure on renal perfusion and function in cases undergoing robotic lower tract urologic surgeries, and to assess the contribution of either mannitol or nitroglycerin infusion to the renal hemodynamic/function alterations during pneumoperitoneum.

ELIGIBILITY:
Inclusion Criteria:

* ASA class I - III
* Normal renal functions or Mild renal disease (GFR < 60 ml/min &/or presence of albuminuria > 30 mg/dl)

Exclusion Criteria:

* BMI > 40
* Previous renal surgery
* Moderate (GFR 30 - 59 mg/dl) & severe (GFR 15 - 29 mg/dl) renal impairment
* Decompensated cardiac disease: New York Heart Association (NYHA) class 3 or 4
* Allergy to mannitol or nitroglycerin

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-05-12 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Cystatin C level | 24 hours
  Serum Cystatin C value in mg/l

CONTACTS AND LOCATIONS:
Overall Officials: Ashgan R Ali, MD, Study Chair — Kasr Al-Ainy Hospital, Faculty of Medicine, Cairo University; Nazmy S Mikhael, MD, Principal Investigator — Kasr Al-Ainy Hospital, Faculty of Medicine, Cairo University; Manar H Mohamed, Study Director — Kasr Al-Ainy Hospital, Faculty of Medicine, Cairo University
Locations (1):
- Cairo University Hospitals, Cairo, Egypt